CLINICAL TRIAL: NCT05962801
Title: Regular Home Use of Dual-light Photodynamic Therapy as an Adjunct to Non-surgical Periodontal Treatment in Smokers
Brief Title: Use of Dual-light Photodynamic Therapy as an Adjunct to Periodontal Treatment in Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Dimitra Sakellari, Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 176/30-11-2022
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Periodontitis; Dual- Light Photodynamic Therapy; Smoking, Cigarette; Non-surgical Periodontal Therapy
Keywords: periodontitis; periodontal diseases; photodynamic therapy; photothermal therapy; smoking; non-surgical periodontitis therapy
MeSH Terms: conditions — Periodontitis; Cigarette Smoking; Periodontal Diseases; Smoking

STUDY DESIGN:
Intervention Model Description: Randomized, controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumoral users (Active Comparator): Use of Lumoral device and Lumorinse mouthwash once per day for 6 months and performance of oral hygiene twice per day for 6 months.
  Interventions: Device: Lumoral device, Lumorinse
- Lumoral non-users (No Intervention): No use of Lumoral device and Lumorinse mouthwash. Performance of oral hygiene twice per day for 6 months.

INTERVENTIONS:
Device: Lumoral device, Lumorinse — Regular use of dual-light photodynamic therapy at home
  Arms: Lumoral users

SUMMARY:
The goal of this controlled clinical trial is to investigate the impact of regular home use of Lumoral device as an adjunct treatment compared to non-surgical periodontitis treatment (NSPT) alone on biofilm removal and host response in Stage III and Grade C smoking periodontitis patients at 6 months.The main question aims to answer is:

• Does regular use of dual-light photodynamic therapy benefit NSPT in Stage III and Grade C smoking periodontitis patients?

30 participants will be asked to use Lumoral device every night before performing oral hygiene for 10 minutes, while the other 30 patients will be asked to perform only oral hygiene. Both of these groups will receive NSPT and will be followed for 6 months from baseline.

DETAILED DESCRIPTION:
The objective of this study is to investigate the impact of regular home use of Lumoral device® as an adjunct treatment compared to non-surgical periodontal treatment alone on biofilm removal and host response in Stage III and Grade C smoking periodontitis patients at 6 months.

Lumoral® is based on a dual-wavelength LED light that activates Lumorinse® (exocellular) and bacteria porphyrins (endocellular), resulting in the formation of reactive oxygen species (ROS). ROS and heat induce a series of photochemical and biological events that cause irreversible inactivation leading to the death of undesired bacteria. This device is designed for home use.

Therefore it is hypothesized that its adjunct use in the treatment of periodontitis could lead to better outcomes compared to traditional periodontal treatment. In order to investigate this impact, clinical and microbiological measurements will be compared between patients who will be treated with conventional non-surgical periodontal treatment and patients who will receive the Lumoral device® as an adjunct to the periodontal treatment. The patients who receive the device will use it every day for four months. Both groups will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal disease Stage III and Grade C with at least 6 sites with probing depth (PD) and clinical attachment loss (CAL) ≥5 mm and bleeding on probing (BoP) ≥15 teeth
* aged ≥35
* Smokers smoking ≥10 cigarettes per day

Exclusion Criteria:

* Patients allergic to indocyanine
* Patients with active carious lesions
* Need for prophylactic antimicrobial coverage
* Scaling and root planing in the previous 6 months
* Non-smoking status or smoking less than 10 cigarettes per day
* Antimicrobial therapy in the previous 6 months
* Immunomodifying conditions/ diseases (e.g. diabetes mellitus, rheumatoid arthritis, osteoporosis)
* Long-term use of medication that could interfere with periodontal response (e.g. biphosphonates)
* Pregnancy or lactation

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in bleeding on probing (BOP) | baseline, 2 weeks, 2 months, 6 months
  Changes in the presence of bleeding when probing at 6 sites per tooth. It is evaluated dichotomously.

SECONDARY OUTCOMES:
Changes of pocket depths | baseline, 2 months, 6 months
  Changes in measurement in millimeters of the depth from the gingival margin to the epithelial attachment in unhealthy gingival tissue at 6 sites per tooth
Changes in clinical attachment level | baseline, 2 months, 6 months
  Changes in measurement of the position of the gingival margin in relation to the cemento-enamel junction (CEJ) at 6 sites per tooth
Difference in the number of "closed" pockets | baseline, 2 months, 6 months
  Differences in the number of pockets with depth≤ 4mm and no BOP between the test and the control group
a-MMP8 saliva concentration | baseline, 2 weeks, 2 months, 6 months
  Periosafe chair-side tests and the ORALyzer (an advanced lateral flow (aLF) reader) are utilized in order to quantify active MMP-8 in subjects' saliva
Changes in Turetsky Modified Quigley-Hein Plaque Index (TMQHPI) | baseline, 2 weeks, 2 months, 6 months
  Changes in TMQHPI in buccal surfaces of the upper and lower anterior teeth.
  A score of 0 to five is assigned to each buccak surface of upper and lower anterior teeth, as follows:
  0 = No plaque.
  1. = Separate flecks of plaque at the cervical margin of the tooth.
  2. = A thin continuous band of plaque (up to one mm) at the cervical margin of the tooth.
  3. = A band of plaque wider than one mm but covering less than one-third of the crown of the tooth.
  4. = Plaque covering at least one-third but less than two thirds of the crown of the tooth.
  5. = Plaque covering two-thirds or more of the crown of the tooth. An index for the anterior teeth is determined by dividing the total score by the number surfaces examined. The score is rounded up to the second decimal number and it ranges from 0 to 5.
Oral health-related quality of life questionnaire (OHQL) | 2 months, 6 months
  OHQL includes the following questions:
  1. Did you use Lumoral® as instructed to you?
  2. Did you find Lumoral® easy to use?
  3. Did you feel any discomfort when using Lumoral®?
  4. Did you discontinue the use of Lumoral® due to this discomfort?
  5. Did Lumoral® help you perform oral hygiene?
  6. Has bad breath been decreased?
  7. Has bleeding of the gums been decreased?
  8. Would you recommend Lumoral®?
  9. Would you buy Lumoral® if its cost was about 200 €?
  All questions will be answered with a 'Yes' or 'No'
Changes in the presence of periopathogens in the deepest pocket | baseline, 2 months, 6 months
  Subgingival plaque sample is collected from the deepest pocket of each patient and the presence of periopathogens is detected

CONTACTS AND LOCATIONS:
Overall Officials: Dimitra Sakellari, Professor, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- Dental School of Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
Patients' data will be recorded in the electronic patients' database of the Dental School of Aristotle University of Thessaloniki and only the researchers of this study will have access to them.

REFERENCES:
- [Background] AlSarhan MA, Altammami MA, Alaqeely RS, AlEbdi A, Jasser RA, Otaibi DA, Oraini SA, Habib SR, Alqahtani L, Alduhaymi IS, Alrabiah DK, Alaradi M, Alyamani EJ. Short-term improvement of clinical parameters and microbial diversity in periodontitis patients following Indocyanine green-based antimicrobial photodynamic therapy: A randomized single-blind split-mouth cohort. Photodiagnosis Photodyn Ther. 2021 Sep;35:102349. doi: 10.1016/j.pdpdt.2021.102349. Epub 2021 May 24. PMID 34033939
- [Background] Lahteenmaki H, Patila T, Raisanen IT, Kankuri E, Tervahartiala T, Sorsa T. Repeated Home-Applied Dual-Light Antibacterial Photodynamic Therapy Can Reduce Plaque Burden, Inflammation, and aMMP-8 in Peri-Implant Disease-A Pilot Study. Curr Issues Mol Biol. 2022 Mar 8;44(3):1273-1283. doi: 10.3390/cimb44030085. PMID 35723308
- [Background] Trujiilo K, Raisanen IT, Sorsa T, Patila T. Repeated Daily Use of Dual-Light Antibacterial Photodynamic Therapy in Periodontal Disease-A Case Report. Dent J (Basel). 2022 Sep 1;10(9):163. doi: 10.3390/dj10090163. PMID 36135158
- [Background] Alassiri S, Parnanen P, Rathnayake N, Johannsen G, Heikkinen AM, Lazzara R, van der Schoor P, van der Schoor JG, Tervahartiala T, Gieselmann D, Sorsa T. The Ability of Quantitative, Specific, and Sensitive Point-of-Care/Chair-Side Oral Fluid Immunotests for aMMP-8 to Detect Periodontal and Peri-Implant Diseases. Dis Markers. 2018 Aug 5;2018:1306396. doi: 10.1155/2018/1306396. eCollection 2018. PMID 30154936
- [Background] Jansson H, Wahlin A, Johansson V, Akerman S, Lundegren N, Isberg PE, Norderyd O. Impact of periodontal disease experience on oral health-related quality of life. J Periodontol. 2014 Mar;85(3):438-45. doi: 10.1902/jop.2013.130188. Epub 2013 Jul 29. PMID 23895254
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Background] Chambrone L, Wang HL, Romanos GE. Antimicrobial photodynamic therapy for the treatment of periodontitis and peri-implantitis: An American Academy of Periodontology best evidence review. J Periodontol. 2018 Jul;89(7):783-803. doi: 10.1902/jop.2017.170172. PMID 30133749
- [Background] Pakarinen S, Saarela RKT, Valimaa H, Heikkinen AM, Kankuri E, Noponen M, Alapulli H, Tervahartiala T, Raisanen IT, Sorsa T, Patila T. Home-Applied Dual-Light Photodynamic Therapy in the Treatment of Stable Chronic Periodontitis (HOPE-CP)-Three-Month Interim Results. Dent J (Basel). 2022 Nov 2;10(11):206. doi: 10.3390/dj10110206. PMID 36354651
- [Derived] Vakaki C, Fragkioudakis I, Patila T, Sakellari D. Regular home use of dual-light photodynamic therapy as an adjunct to non-surgical periodontal treatment in smokers: a single-center randomized controlled clinical trial. Clin Oral Investig. 2025 Nov 6;29(12):553. doi: 10.1007/s00784-025-06600-1. PMID 41196397

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT05962801/Prot_SAP_001.pdf